CLINICAL TRIAL: NCT02673307
Title: Chewing Gum and Gastric Emptying of Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lionel Bouvet (Other)
Responsible Party: Sponsor-Investigator, Lionel Bouvet, MD, PhD, Hôpital Edouard Herriot
Organization: Hôpital Edouard Herriot (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-A00009-42; L15-206 (Other: Comité de Protection des Personnes Sud Est IV)
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Comparison of Gastric Emptying Rate of Water When Chewing Gum or Not

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Controle (No Intervention): The volunteer does not chew gum during the study period
- Chewing gum (Experimental): The volunteer chews gum during the first 45 min after ingestion of 250 ml water
  Interventions: Behavioral: 1 chewing gum over 45 minutes

INTERVENTIONS:
Behavioral: 1 chewing gum over 45 minutes
  Arms: Chewing gum

SUMMARY:
The aims of this prospective cross over study was to compare the gastric emptying of 250 ml water in fasting volunteers, in two situations : without chewing gum or while chewing gum during 45 min

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2 volunteers

Exclusion Criteria:

* digestive diseases, gastroparesis
* Smokers
* Pregnancy
* Diabetes Mellitus
* Medication affecting gastric motility
* Previous gastrointestinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the rate of gastric emptying of 250 ml water when chewing or not chewing gum, as assessed by the ultrasound measurement of antral area performed each 20 min | every 20 minutes during 120 min

CONTACTS AND LOCATIONS:
Overall Officials: Lionel BOUVET, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Femme Mère Enfant - Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Derived] Bouvet L, Loubradou E, Desgranges FP, Chassard D. Effect of gum chewing on gastric volume and emptying: a prospective randomized crossover study. Br J Anaesth. 2017 Nov 1;119(5):928-933. doi: 10.1093/bja/aex270. PMID 29077816